CLINICAL TRIAL: NCT01696734
Title: Treatment Protocol for the Compassionate Use of Domperidone
Brief Title: Domperidone in Treating Patients With Gastrointestinal Disorders
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2012-0261; NCI-2012-02093 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2012-0261 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2012-09-27; First posted 2012-10-01 (Estimated); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Digestive System Disorder; Dyspepsia; Esophagitis; Gastroesophageal Reflux Disease; Gastroparesis; Heartburn; Nausea and Vomiting
MeSH Terms: conditions — Digestive System Diseases; Dyspepsia; Esophagitis; Gastroesophageal Reflux; Gastroparesis; Heartburn; Nausea; Vomiting | interventions — Domperidone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (domperidone) (Experimental): Patients receive domperidone PO TID or QID. Treatment continues in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Domperidone; Other: Questionnaire Administration

INTERVENTIONS:
Drug: Domperidone — Given PO
  Other Names: KW 5338; Motilium; R 33,812
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This phase III trial studies how well domperidone works in treating patients with gastrointestinal disorders. Domperidone may help control chronic gastrointestinal disorders and their symptoms, such as pain, bloating, and nausea and vomiting, by stimulating contraction of the stomach to increase its ability to empty itself of food.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To provide treatment with domperidone to patients >= 16 years of age where, according to the investigators' judgment, a prokinetic effect is needed for the relief of gastrointestinal (GI) motility disorders.

OUTLINE:

Patients receive domperidone orally (PO) thrice daily (TID) or four times daily (QID). Treatment continues in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for at least 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Patients with GI disorders who have failed standard therapy
* Symptoms or manifestations of: a) gastroparesis; b) refractory gastroesophageal reflux disease (GERD) including persistent esophagitis, refractory heartburn, reflux-related laryngitis, and respiratory symptoms; or c) severe dyspepsia
* Completion of a comprehensive evaluation, including clinical history and physical examination, to eliminate other causes of their symptoms
* Patient has signed the informed consent document agreeing to the use of the study drug, domperidone
* White blood cell (WBC) with differential greater than 3,000/ml
* Alkaline phosphatase less than 1.5 x upper limit of normal
* Alanine aminotransferase (ALT) less than 2 x upper limit of normal
* Aspartate aminotransferase (AST) less than 2 x upper limit of normal
* Bilirubin less than or equal to 2 x upper limit of normal
* Blood urea nitrogen (BUN) less than 2 x upper limit of normal
* Creatinine less than 1.5 x upper limit of normal
* Stable hemoglobin greater than or equal to 8.0 g/dl
* Potassium between range of 3.0 to 5.5
* Magnesium level between 1.6-2.6 mg

Exclusion Criteria:

* Patients with the following cardiac diagnoses: ventricular tachycardia or fibrillation; Torsade des Pointes; clinically significant bradycardia; sinus node dysfunction; heart block; prolonged QTc interval (QTc > 450 milliseconds for males, QTc > 470 milliseconds for females); prior specific cardiovascular conditions of clinically significant valvular heart disease requiring medication, ischemic, or pulmonary heart disease; cardiomyopathy; history of heart failure
* Patients who are receiving antiarrhythmic medications with action on repolarization times (with prolongation of the QTc interval such as amiodarone, disopyramide, dofetilide, flecainide, ibutilide, quinidine, sotalol, dronedarone etc.)
* Patients who are receiving monoamine oxidase (MAO) inhibitors
* Patients with a history of or active liver failure
* Clinically significant electrolyte disorders including sodium < 130 or > 145 and/or potassium < 3.0 or > 5.5 and/or magnesium < 1.6 or > 2.6
* GI hemorrhage or obstruction experienced within the previous 6 weeks
* Presence of a prolactinoma (prolactin-releasing pituitary tumor)
* Pregnant or breast-feeding female (women of childbearing potential [WOCBP], defined as not post-menopausal for 12 months or without previous surgical sterilization, must have a negative urine pregnancy test within 30 days of the first administration of domperidone and must either commit to continued abstinence from heterosexual intercourse or use an effective method of birth control during the course of the study)
* Known allergy to domperidone

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2012-10-23 (Actual); Primary Completion 2027-10-31 (Estimated); Study Completion 2027-10-31 (Estimated)

PRIMARY OUTCOMES:
Attenuation of symptoms associated with disorder(s) of gastrointestinal motility, measured by change in Gastroparesis Cardinal Symptom Index (GSCI) score from baseline | Baseline to 8 weeks
  Scale ranges from "0" meaning "None" to "5" meaning "Very Severe".
  Patients will be classified as either "new" or "continuing" at the baseline visit. A new patient will have a "response" if he/she has a 25% reduction in GCSI at 8 weeks. A continuing patient will already have early benefit to treatment so will have a "response" if the GCSI score does not increase more than 20% over baseline at 8 weeks. Summary statistics including number (n), mean, standard deviation, median, minimum, and maximum will be computed. Bayesian 95% credible intervals will be computed.

SECONDARY OUTCOMES:
Change in patients' self-report of symptoms | Baseline to 30 days after completion of study treatment
  Summary statistics including n, mean, standard deviation, median, minimum, and maximum will be computed. Bayesian 95% credible intervals will be computed.
Incidence of toxicities assessed according to the Common Terminology Criteria for Adverse Events version 4.0 | Up to 30 days after completion of study treatment
  Summary statistics including n, mean, standard deviation, median, minimum, and maximum will be computed. Bayesian 95% credible intervals will be computed. Patient adverse events will be tabulated by symptom, grade, and relationship to study drug.

CONTACTS AND LOCATIONS:
Overall Officials: Mehnaz Shafi, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org